CLINICAL TRIAL: NCT05575219
Title: Protocolized Initiation of Clonidine to Prevent Dexmedetomidine Withdrawal: A Prospective Cohort Study
Brief Title: Protocolized Initiation of Clonidine to Prevent Dexmedetomidine Withdrawal
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Andrea Leigh Heifner, Clinical Fellow, The University of Texas Health Science Center, Houston
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HSC-MS-22-0410
Record Dates: First submitted 2022-10-05; First posted 2022-10-12 (Actual); Results first posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Withdrawal; Therapeutic Substance
MeSH Terms: interventions — Clonidine; clonidine 4-methylisothiocyanate

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Usual care (without protocolized clonidine initiation) (Active Comparator): Participants will be observed for dexmedetomidine withdrawal and clonidine will be started at clinician discretion.
  Interventions: Drug: Clonidine (without protocolized initiation)
- Intervention (protocolized clonidine initiation) (Experimental): A protocol for clonidine initiation will be implemented based on the time on dexmedetomidine and the average hourly dose of dexmedetomidine.
  Interventions: Drug: Clonidine (protocolized initiation)

INTERVENTIONS:
Drug: Clonidine (without protocolized initiation) — Participants will be observed for dexmedetomidine withdrawal and clonidine will be started at clinician discretion.
  Other Names: Clondine
  Arms: Usual care (without protocolized clonidine initiation)
Drug: Clonidine (protocolized initiation) — * Observe participants without initiating clonidine with dexmedetomidine infusion time of 72-119 hours. To wean off dexmedetomidine, decrease the infusion by 25% of the starting dose every 6 hours.
  * Begin clonidine at 1 mcg/kg enterally every 6 hours for participants with dexmedetomidine infusion time of 120-144 hours.
  * Begin clonidine at 1.5 mcg/kg enterally every 6 hours for participants with dexmedetomidine infusion times of 145-167 hours.
  * Begin clonidine at 2 mcg/kg enterally every 6 hours for participants with dexmedetomidine infusion time of >/= 168 hours or with infusion time of 120-167 hours at doses >/= 1.1 mcg/kg/min.
  * If clonidine is started decrease the dexmedetomidine infusion by 25% of the starting dose 1 hour after each dose of clonidine until off (wean every 6 hours).
  Other Names: Clondine
  Arms: Intervention (protocolized clonidine initiation)

SUMMARY:
The purpose of this study is to determine if the protocolized use of clonidine will reduce dexmedetomidine withdrawal symptoms, reduce PICU length of stay, and reduce costs related to sedation during hospital admission.

ELIGIBILITY:
Inclusion Criteria:

* Dexmedetomidine infusion for greater than or equal to 72 hours

Exclusion Criteria:

* Admission for head trauma
* Psychiatric history
* Use of alpha-2 agonist medications at home
* Death while on dexmedetomidine

Ages: 4 Weeks to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 128 (Actual)
Dates: Start 2022-10-08 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Heifner, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Children's Memorial Hermann Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berkenbosch JW. Dexmedetomidine and pediatric (cardiac) critical care--are we there yet? Pediatr Crit Care Med. 2010 Jan;11(1):148-9. doi: 10.1097/PCC.0b013e3181bc57c0. No abstract available. PMID 20051795
- [Background] Berrens ZJ, Sauro AL, Tillman EM. Prevention of Withdrawal in Pediatric Patients Receiving Long-term Dexmedetomidine Infusions. J Pediatr Pharmacol Ther. 2021;26(1):81-86. doi: 10.5863/1551-6776-26.1.81. Epub 2021 Jan 4. PMID 33424504
- [Background] Bhatt K, Thompson Quan A, Baumgartner L, Jia S, Croci R, Puntillo K, Ramsay J, Bouajram RH. Effects of a Clonidine Taper on Dexmedetomidine Use and Withdrawal in Adult Critically Ill Patients-A Pilot Study. Crit Care Explor. 2020 Nov 3;2(11):e0245. doi: 10.1097/CCE.0000000000000245. eCollection 2020 Nov. PMID 33163969
- [Background] Curley MA, Harris SK, Fraser KA, Johnson RA, Arnold JH. State Behavioral Scale: a sedation assessment instrument for infants and young children supported on mechanical ventilation. Pediatr Crit Care Med. 2006 Mar;7(2):107-14. doi: 10.1097/01.PCC.0000200955.40962.38. PMID 16446601
- [Background] Darnell C, Steiner J, Szmuk P, Sheeran P. Withdrawal from multiple sedative agent therapy in an infant: is dexmedetomidine the cause or the cure? Pediatr Crit Care Med. 2010 Jan;11(1):e1-3. doi: 10.1097/PCC.0b013e3181a66131. PMID 20051785
- [Background] Franck LS, Harris SK, Soetenga DJ, Amling JK, Curley MA. The Withdrawal Assessment Tool-1 (WAT-1): an assessment instrument for monitoring opioid and benzodiazepine withdrawal symptoms in pediatric patients. Pediatr Crit Care Med. 2008 Nov;9(6):573-80. doi: 10.1097/PCC.0b013e31818c8328. PMID 18838937
- [Background] Franck LS, Scoppettuolo LA, Wypij D, Curley MAQ. Validity and generalizability of the Withdrawal Assessment Tool-1 (WAT-1) for monitoring iatrogenic withdrawal syndrome in pediatric patients. Pain. 2012 Jan;153(1):142-148. doi: 10.1016/j.pain.2011.10.003. Epub 2011 Nov 16. PMID 22093817
- [Background] Haenecour AS, Seto W, Urbain CM, Stephens D, Laussen PC, Balit CR. Prolonged Dexmedetomidine Infusion and Drug Withdrawal In Critically Ill Children. J Pediatr Pharmacol Ther. 2017 Nov-Dec;22(6):453-460. doi: 10.5863/1551-6776-22.6.453. PMID 29290746
- [Background] Lardieri AB, Fusco NM, Simone S, Walker LK, Morgan JA, Parbuoni KA. Effects of Clonidine on Withdrawal From Long-term Dexmedetomidine in the Pediatric Patient. J Pediatr Pharmacol Ther. 2015 Jan-Feb;20(1):45-53. doi: 10.5863/1551-6776-20.1.45. PMID 25859170
- [Background] Liu J, Miller J, Ferguson M, Bagwell S, Bourque J. The Impact of a Clonidine Transition Protocol on Dexmedetomidine Withdrawal in Critically Ill Pediatric Patients. J Pediatr Pharmacol Ther. 2020;25(4):278-287. doi: 10.5863/1551-6776-25.4.278. PMID 32461740
- [Background] Nguyen TL, Lam WM, Orr H, Gulbis B, Mauricio R, Tom E, Modem VM, Coronado-Munoz A. Clonidine for the Treatment of Agitation After Dexmedetomidine Discontinuation in Pediatric Patients: A Retrospective Cohort Study. J Pediatr Pharmacol Ther. 2021;26(8):821-827. doi: 10.5863/1551-6776-26.8.821. Epub 2021 Nov 10. PMID 34790072
- [Background] Shutes BL, Gee SW, Sargel CL, Fink KA, Tobias JD. Dexmedetomidine as Single Continuous Sedative During Noninvasive Ventilation: Typical Usage, Hemodynamic Effects, and Withdrawal. Pediatr Crit Care Med. 2018 Apr;19(4):287-297. doi: 10.1097/PCC.0000000000001451. PMID 29341985
- [Background] Thompson RZ, Gardner BM, Autry EB, Day SB, Krishna AS. Survey of the Current Use of Dexmedetomidine and Management of Withdrawal Symptoms in Critically Ill Children. J Pediatr Pharmacol Ther. 2019 Jan-Feb;24(1):16-21. doi: 10.5863/1551-6776-24.1.16. PMID 30837809
- [Background] Traube C, Silver G, Kearney J, Patel A, Atkinson TM, Yoon MJ, Halpert S, Augenstein J, Sickles LE, Li C, Greenwald B. Cornell Assessment of Pediatric Delirium: a valid, rapid, observational tool for screening delirium in the PICU*. Crit Care Med. 2014 Mar;42(3):656-63. doi: 10.1097/CCM.0b013e3182a66b76. PMID 24145848
- [Background] Weber MD, Thammasitboon S, Rosen DA. Acute discontinuation syndrome from dexmedetomidine after protracted use in a pediatric patient. Paediatr Anaesth. 2008 Jan;18(1):87-8. doi: 10.1111/j.1460-9592.2007.02377.x. No abstract available. PMID 18095980
- [Background] Lee MM, Caylor K, Gockenbach N. Evaluating the Transition From Dexmedetomidine to Clonidine for the Prevention of Withdrawal in Critically Ill Pediatric Patients. J Pediatr Pharmacol Ther. 2020;25(2):104-110. doi: 10.5863/1551-6776-25.2.104. PMID 32071584
- [Background] Miller JL, Allen C, Johnson PN. Neurologic withdrawal symptoms following abrupt discontinuation of a prolonged dexmedetomidine infusion in a child. J Pediatr Pharmacol Ther. 2010 Jan;15(1):38-42. PMID 22477791

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention (Protocolized Clonidine Initiation): A protocol for clonidine initiation will be implemented based on the time on dexmedetomidine and the average hourly dose of dexmedetomidine.
  Clonidine (protocolized initiation): - Observe participants without initiating clonidine with dexmedetomidine infusion time of 72-119 hours. To wean off dexmedetomidine, decrease the infusion by 25% of the starting dose every 6 hours.
  * Begin clonidine at 1 mcg/kg enterally every 6 hours for participants with dexmedetomidine infusion time of 120-144 hours.
  * Begin clonidine at 1.5 mcg/kg enterally every 6 hours for participants with dexmedetomidine infusion times of 145-167 hours.
  * Begin clonidine at 2 mcg/kg enterally every 6 hours for participants with dexmedetomidine infusion time of >/= 168 hours or with infusion time of 120-167 hours at doses >/= 1.1 mcg/kg/min.
  * If clonidine is started decrease the dexmedetomidine infusion by 25% of the starting dose 1 hour after each dose of clonidine until off (wean every 6 hours).
Period: Overall Study
Arm/Group | Usual Care (Without Protocolized Clonidine Initiation) | Intervention (Protocolized Clonidine Initiation)
Started | 96 | 32
Completed | 96 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care (Without Protocolized Clonidine Initiation) | Intervention (Protocolized Clonidine Initiation) | Total
Number analyzed (Participants) | 96 | 32 | 128
Age, Continuous [Median (Inter-Quartile Range); unit: months] | 10 [3 to 28.5] | 16.5 [4.75 to 113.75] | 10.5 [3.75 to 47.75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 21 | 75
  Male | 42 | 11 | 53
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 96 | 32 | 128
Weight [Median (Inter-Quartile Range); unit: kilograms] | 7.515 [4.525 to 12.325] | 10.95 [5.885 to 26.475] | 8.418 [4.778 to 16.5]
Primary Diagnosis [Count of Participants; unit: Participants]
  Cardiac Diagnosis | 40 | 0 | 40
  Respiratory Diagnosis | 45 | 22 | 67
  Neurologic Diagnosis | 3 | 2 | 5
  Sepsis Diagnosis | 4 | 2 | 6
  Hematology/Oncology Diagnosis | 2 | 2 | 4
  Other Diagnosis | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Withdrawal
Description: The number of participants with withdrawal is reported. Withdrawal is defined as: (increase in heart rate, systolic blood pressure, and/or diastolic blood pressure by at least 10% from the 24 hours prior to dexmedetomidine weaning to the 24 hours after dexmedetomidine is discontinued) AND (two documented WAT (Withdrawal assessment tool)-1 scores of ≥ 3 and/or two study questionnaire scores of ≥ 3). WAT and questionnaire scores will be collected every 12 hours starting with the first dexmedetomidine wean until 72 hours after dexmedetomidine is discontinued.
  WAT-1 is a scoring tool used to evaluate symptoms of withdrawal with a total score that ranges from 0 to 12. The higher the score the more severe the withdrawal.
  The study questionnaire is used to evaluate degree of agitation and/or insomnia with a total score that ranges from 0 to 7, a higher score indicates higher degrees of agitation and/or insomnia.
Time Frame: from the time dexmedetomidine is first weaned until 72 hours after dexmedetomidine is off (about 3-14 days)
Population: Data were not collected from 5 participants in the Usual care (without protocolized clonidine initiation) arm. Data were not collected from 2 participants in the Intervention (protocolized clonidine initiation) arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care (Without Protocolized Clonidine Initiation) | Intervention (Protocolized Clonidine Initiation)
Number analyzed (Participants) | 91 | 30
Participants | 33 | 10

2. Secondary Outcome: Hours on Dexmedetomidine
Description: number of total hours on dexmedetomidine
Time Frame: During time in Pediatric Intensive Care Unit (about 260 Hours)
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Usual Care (Without Protocolized Clonidine Initiation) | Intervention (Protocolized Clonidine Initiation)
Number analyzed (Participants) | 96 | 32
Hours | 153.43 [114.79 to 218.62] | 155.33 [132.83 to 260.23]

3. Secondary Outcome: Pediatric Intensive Care Unit (PICU) Length of Stay
Description: number of days in the PICU
Time Frame: During time in Pediatric Intensive Care Unit (about 10 to 30 days)
Population: Data were not collected for 8 participants in the Usual care (without protocolized clonidine initiation) arm.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Usual Care (Without Protocolized Clonidine Initiation) | Intervention (Protocolized Clonidine Initiation)
Number analyzed (Participants) | 88 | 32
Days | 13 [9 to 28] | 10.5 [8.75 to 16.25]

4. Secondary Outcome: Dexmedetomidine Cost Per Kilogram During Hospitalization
Time Frame: During time in Pediatric Intensive Care Unit (about 24 days)
Measure: Median (Inter-Quartile Range); unit: dollars per kilogram
Arm/Group | Usual Care (Without Protocolized Clonidine Initiation) | Intervention (Protocolized Clonidine Initiation)
Number analyzed (Participants) | 96 | 32
dollars per kilogram | 19.98 [14.5 to 32.72] | 29.46 [20.19 to 47.64]

5. Secondary Outcome: Clonidine Cost Per Kilogram During Hospitalization
Time Frame: During time in Pediatric Intensive Care Unit (about 24 days)
Measure: Median (Inter-Quartile Range); unit: cents per kilogram
Arm/Group | Usual Care (Without Protocolized Clonidine Initiation) | Intervention (Protocolized Clonidine Initiation)
Number analyzed (Participants) | 96 | 32
cents per kilogram | 0.06 [0.03 to 0.14] | 0.05 [0.02 to 0.1]

ADVERSE EVENTS:
Time Frame: From baseline to time in PICU (about 24 days)
Arm/Group | Usual Care (Without Protocolized Clonidine Initiation) | Intervention (Protocolized Clonidine Initiation)
All-Cause Mortality (participants affected / at risk) | 0/96 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/96 | 0/32
Other Adverse Events (participants affected / at risk) | 0/96 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-15): https://cdn.clinicaltrials.gov/large-docs/19/NCT05575219/Prot_SAP_000.pdf